CLINICAL TRIAL: NCT04461951
Title: Exploring the Relationship Between Nutrition, gUT Microbiota, and BRain AgINg in Community-dwelling Seniors: the NutBrain Study
Brief Title: Nutrition, gUT Microbiota, and BRain AgINg: the NutBrain Study
Acronym: NutBrain
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: IRCCS National Neurological Institute "C. Mondino" Foundation (Other)
Collaborators: Institute of Biomedical Technologies-National Research Council (ITB-CNR) (Unknown)
Responsible Party: Sponsor
Other Study IDs: NutBrain2018
Record Dates: First submitted 2020-06-29; First posted 2020-07-08 (Actual); Last update posted 2020-07-08 (Actual); Status verified 2020-07

CONDITIONS: Cognitive Dysfunction; Dietary Habits
Keywords: Cognitive Impairments, Dietary habits, Gut Microbiota, Brain
MeSH Terms: conditions — Cognitive Dysfunction; Feeding Behavior

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Blood and stool samples are collected from each participant and stored in the biorepository at the Hospital for gut microbiota analysis and the evaluation of putative biological markers.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Community dwelling seniors: Participants are visited at the research facility in their residence town by a trained team. Informed consent form is completed at the research facility prior to data collection. In those individuals without capacity to give full informed consent, proxy consent is collected from relatives or caregivers. This 2-hours interview includes a face-to-face administration of a neuropsychological battery of tests and questionnaires to inquire about socio-demographic, occupational, and social-economic data, education, medical conditions and drug use, lifestyle habits, functional status, and dietary behaviours.
  Interventions: Other: Lifestyles (exposure)

INTERVENTIONS:
Other: Lifestyles (exposure) — no intervention
  Other Names: no intervention

SUMMARY:
Epidemiological evidence suggests that healthy diet is associated with a slowdown of cognitive decline leading to dementia, but the underlying mechanisms are still partially unexplored. Diet is the main determinant of gut microbiota' composition, which in turn impacts on brain structures and functions, however to date no studies on this topic are available. The goal of the present paper is to describe the design and methodology of the NutBrain Study aimed at investigating the association of dietary habits with cognitive function, and their role in modulating the gut microbiota composition, and brain measures as well.

This is a population-based cohort study of community-dwelling adults aged 65 years or more living in Northern Milan, Italy. At the point of presentation people are screened for cognitive functions. Socio-demographic characteristics along with lifestyles and dietary habits, medical history, drugs, functional status, and anthropometric measurements are also recorded. Individuals suspected to have cognitive impairment at the screening phase undergo a clinical evaluation including a neurological examination and a Magnetic Resonance Imaging (MRI) scanning (both structural and functional). Stool and blood samples for the gut microbiota analysis and for the evaluation of putative biological markers are also collected. For each subject with a confirmed diagnosis of Mild Cognitive Impairment (MCI), two cognitively intact controls of the same sex and age are visited. The investigators intend to enrol at least 683 individuals for the screening phase and approximately 240 persons for the clinical assessment.

The NutBrain is an innovative study that incorporates modern and advanced technologies (i.e. microbiome and neuroimaging) into traditional epidemiologic design. The study represents a unique opportunity to address key questions about the role of modifiable risk factors on cognitive impairment, with a particular focus on dietary habits and their association with gut microbiota and markers of the brain-aging process. These findings will help to encourage and plan lifestyle interventions, for both prevention and treatment, aiming at promoting healthy cognitive ageing.

DETAILED DESCRIPTION:
The NutBrain Study aims to understand the biological mechanisms through which diet influences cognitive disorders with a special focus on the impact of nutrition on gut microbiota and brain characteristics, by applying a novel multi-level approach that integrates traditional epidemiological methods with neuroimaging and gut microbiota profiling. Aims of the NutBrain study are: i) to estimate the occurrence of MCI and other cognitive disorders in community-dwelling older people aged 65 + years; ii) to investigate the association between lifestyle habits and cognitive ageing outcomes; iii) to explore the role of diet, in modulating the gut microbiota composition, which in turn impacts on brain structures and functions as well.

The NutBrain Study is an ongoing population-based cohort study promoted by the Institute of Biomedical Technologies of the National Research Council (ITB-CNR, Segrate, Italy) and the Hospital IRCCS Fondazione Mondino (Pavia, Italy). The NutBrain Study is structured in three phases:

T=1 Participant's recruitment. The study is performed in two sites in the outskirt of North-Milan: Bollate and Baranzate. A random sample is drawn from the official register of residents in the two municipalities. Inclusion criteria are: attending a medical appointment in the research facility, living at home in one of the two municipalities, and being 65+ years. Eligible population is contacted by means of a letter of invitation, in which people are invited to contact the ITB-CNR by phone to schedule the first visit during which he/she is asked to bring last instrumental and clinical exams prescribed by their general practitioner. A comprehensive communication campaign is implemented to publicize and promote the project as well as to foster recruitment. To ensure a high enrolment rate, the Mayors of the two municipalities have been actively involved since the earliest planning stages of the recruitment and have granted patronage to the project. Additionally, the study is promoted and advertised at the community level through different channels: by printing brochures and setting posters in senior recreation centres, shops, pharmacies, medical doctors office, and patients associations; by articles and advertisements in local newspapers, institution websites, as well as in social media (e.g. Facebook, https://www.facebook.com/TheNutBrainStudy/). The NutBrain Study has a website (www.nutbrain.it) where potential participants are directed for further information and can register interest to participate. In addition, to raise awareness, several public events describing the objectives of the proposed study are organized for recruiting eligible people.

T=2 Screening evaluation. Participants are visited at the research facility in their residence town (arranging home visits for disabled individuals) by a trained team. Informed consent form is completed at the research facility prior to data collection. In those individuals without capacity to give full informed consent, proxy consent is collected from relatives or caregivers. This 2-hours interview includes a face-to-face administration of a neuropsychological battery of tests and questionnaires to inquire about socio-demographic, occupational, and social-economic data, education, medical conditions and drug use, lifestyle habits, functional status, and dietary behaviours. At the end of the visit, a stool sampling kit, consisting of a sterile faeces container with instructions explaining the procedure for the stool sample collection, and a 3-day food diary is provided to each participant. The first visit serves to screen each participant for cognitive functions and for identifying inclusion/exclusion criteria in a more comprehensive manner.

T=3 Clinical evaluation. Individuals suspected to have cognitive impairment at the screening neuropsychological tests undergo a clinical examination. Participants are transported from their own home to the Hospital using a private transport service, whose cost is covered entirely by the study. The hospital visit includes a standard neurological examination performed by a neurologist and a 3T Magnetic Resonance Imaging (MRI) scanning. At this stage, blood and stool samples are collected from each participant and stored in the biorepository at the Hospital until processing. For each subject with a clinical diagnosis of MCI, two cognitively intact controls of the same sex and of the closest date of birth are enrolled and visited at the Hospital (case-control design), undergoing the same protocol as MCI individuals.

Date security Data are handled, monitored, computerised, and stored in accordance with the European General Data Protection Regulation (EU) 2016/679 (GDPR) (https://gdpr-info.eu/). All study records, including the consent forms, are kept in a locked filing cabinet at the ITB-CNR where the file server for data storage is located. The file server is firewalled within the ITB-CNR intranet. For privacy and security, a password granted only to the server administrator is required to access to the database. The data forms are double checked for missing data and inconsistencies. Quality of the database entered data is monitored by checking entry for a random sample of participants. Data transfer is protected by means of crypting/decrypting policy and password protection. In the final dataset a unique key identifies each subject to guarantee anonymity. Personal data are regarded as strictly confidential and removed before the exportation procedure. Security of data is guarantee via automatic backups.

ELIGIBILITY:
Inclusion Criteria:

* attending a medical appointment in the research facility
* living at home in one of the two municipalities
* being 65+ years

Exclusion Criteria:

i) neuropsychological criteria:

* subject with dementia, pre-existing cognitive impairment (e.g. aphasia, neglect), concomitant severe psychiatric disease, others neurological conditions (e.g. severe depression and behavioral disorders)
* severe sensory disturbances (e.g. auditory and/or visual loss) that do not allow completing neuropsychological assessment

ii) microbiota' analysis protocol:

* individuals with artificial nutrition in progress
* history of active uncontrolled gastrointestinal disorders or diseases (inflammatory bowel disease, ulcerative colitis, and Crohn's disease)
* subjects who underwent previous major surgery on the gastro-enteric tract, with the exception of cholecystectomy and appendectomy, in the past five years
* use of antibiotics or large doses of commercial probiotics in the 4 weeks prior the visit
* subjects under radio-chemo-therapy

iii) MRI scanning protocol:

* subjects with metal fragments in the body, surgically implanted devices containing metal
* severe claustrophobia
* inability to lie down in the MRI scanner for the duration of the study

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: This is a population-based cohort study of community-dwelling adults aged 65 years or more living in Northern Milan, Italy (Bollate and Baranzate municipalities). A random sample is drawn from the official register of residents in the two municipalities. Eligible population is contacted by means of a letter of invitation, in which people are invited to contact the ITB-CNR by phone to schedule the first visit during which he/she is asked to bring last instrumental and clinical exams prescribed by their general practitioner.
Sampling Method: Probability Sample
Enrollment: 643 (Estimated)
Dates: Start 2019-04-01 (Actual); Primary Completion 2021-10 (Estimated); Study Completion 2022-04 (Estimated)

PRIMARY OUTCOMES:
Number of participants with Mild Cognitive Impairment (MCI) in community dwelling older adults | Screening evaluation at T=2 (24 months after T=0)
  Measured using a battery of well-established neuropsychological tests exploring global cognitive function (Mini Mental State Examination-MMSE) and different cognitive domains: memory (Free and Cues Selective Reminding Test (FCSRT), Logical memory test - Babcock Test, the Rey-Osterrieth Complex Figure Test (ROCF) - delay recall, executive function (Frontal Assessment Battery (FAB)), phonemic and semantic verbal fluency, Trial Making Test (TMT), language (Picture Naming Test), visuo-spatial abilities (Rey-Osterrieth Complex Figure Test (ROCF) - copy). All the test scores are corrected for age, sex, and education and compared with the values available for the Italian population. Diagnosis follows the Albert criteria.

SECONDARY OUTCOMES:
Brain MRI measures | Clinical evaluation at T=3 (32 months after T=0)
  Neuroimaging data are acquired, pre-processed and analyzed at the Hospital. MRI data are acquired using a 3 Tesla Skyra scanner (Siemens, Erlangen, Germany). MRI measures include structural (high resolution T1 anatomical scan - grey matter volume/density, cortical thickness; Diffusion Tensor Imaging scan: white matter microstructural integrity) and functional characteristics (resting state fMRI sequence: functional connectivity at rest)
Bacterial composition of stool samples in terms of relative abundance | Clinical evaluation at T=3 (32 months after T=0)
  Total bacterial DNA is extracted from stool samples and the V3-V4 regions of the microbial 16S rRNA gene are PCR-amplified. Alpha-diversity (i.e.: species diversity within samples) is calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Federica Prinelli, PhD, Principal Investigator — IRCCS C. Mondino Foundation
Locations (1):
- Struttura Semplice Neuropsicologia Clinica/ Centro UVA, Pavia, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Prinelli F, Mastropietro A, Bernini S, Camboni T, Consolandi C, Conti S, Costa A, Cotta Ramusino M, Jesuthasan N, Pansarasa O, Perdixi E, Pichiecchio A, Rizzo G, Scarian E, Severgnini M; NutBrain Study Working Group. Impacts of an antioxidant-rich diet and lifestyle factors on gut microbiota diversity and brain health: An exploratory analysis from the NutBrain study. Clin Nutr. 2026 Feb 2;58:106585. doi: 10.1016/j.clnu.2026.106585. Online ahead of print. PMID 41666842
- [Derived] Perdixi E, Cotta Ramusino M, Costa A, Bernini S, Conti S, Jesuthasan N, Severgnini M, Prinelli F; NutBrain Study Group. Polypharmacy, drug-drug interactions, anticholinergic burden and cognitive outcomes: a snapshot from a community-dwelling sample of older men and women in northern Italy. Eur J Ageing. 2024 Mar 29;21(1):11. doi: 10.1007/s10433-024-00806-0. PMID 38551689
- [Derived] Bernini S, Conti S, Perdixi E, Jesuthasan N, Costa A, Severgnini M, Ramusino MC, Prinelli F; NutBrain Study Group. Investigating the individual and joint effects of socioeconomic status and lifestyle factors on mild cognitive impairment in older Italians living independently in the community: results from the NutBrain study. J Nutr Health Aging. 2024 Mar;28(3):100040. doi: 10.1016/j.jnha.2024.100040. Epub 2024 Jan 26. PMID 38280834
- [Derived] Perdixi E, Bernini S, Conti S, Jesuthasan N, Cotta Ramusino M, Costa A, Prinelli F. Pre-existing mental health disorders and fear of COVID-19 pandemic: Data from a phone survey in community-dwelling older adults recruited in the NutBrain study. Front Psychiatry. 2022 Nov 7;13:995308. doi: 10.3389/fpsyt.2022.995308. eCollection 2022. PMID 36419980
- [Derived] Prinelli F, Jesuthasan N, Severgnini M, Musicco M, Adorni F, Correa Leite ML, Crespi C, Bernini S. Exploring the relationship between Nutrition, gUT microbiota, and BRain AgINg in community-dwelling seniors: the Italian NutBrain population-based cohort study protocol. BMC Geriatr. 2020 Jul 23;20(1):253. doi: 10.1186/s12877-020-01652-2. PMID 32703186
- See also: Official web-site of the NutBrain study project — http://www.nutbrain.it/